CLINICAL TRIAL: NCT02977975
Title: A Randomized Controlled Clinical Trial to Investigate the Efficacy of Traditionally Fermented Sauerkraut in the Treatment of Irritable Bowel Syndrome
Brief Title: Lacto-fermented Sauerkraut in the Treatment of Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Eirik Garnås, Public Health Nutritionist, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016/1130/REK
Record Dates: First submitted 2016-11-26; First posted 2016-11-30 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome; The human microbiome; Microbiota; Gut microbiota; Probiotics; Sauerkraut
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Raw sauerkraut (Experimental): 75 grams of raw, traditionally produced, lacto-fermented sauerkraut, each day for 6 weeks.
  Interventions: Other: Raw sauerkraut
- Pasteurized sauerkraut (Other): 75 grams of pasteurized sauerkraut, each day for 6 weeks.
  Interventions: Other: Pasteurized sauerkraut

INTERVENTIONS:
Other: Raw sauerkraut — Sauerkraut fermentations have been shown to contain a broad range of microorganisms, including Leuconostoc mesenteroides, Lactobacillus plantarum, Leuconostoc citreum, Leuconostoc argentinum, Lactobacillus paraplantarum, and Lactobacillus coryniformis. Some of these bacteria, such as Lactobacillus plantarum, are classified as probiotics.
  Arms: Raw sauerkraut
Other: Pasteurized sauerkraut — Sauerkraut without live bacteria.
  Arms: Pasteurized sauerkraut

SUMMARY:
The aim of the present study is to assess the efficacy of traditionally fermented sauerkraut in the treatment of irritable bowel syndrome.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a chronic gastrointestinal (GI) disorder that affects around 11% of the population globally. Several factors have been implicated in the pathogenesis of IBS, including psychological stress, gastrointestinal motility, and diet . More recently, it has become clear that the gastrointestinal microbiota may play a critical role in the pathophysiology of this functional GI condition.

Several studies have shown that an altered gut microbiota profile is present in at least some subgroups of IBS patients. This may, in part, explain why a proportion of IBS patients have elevated levels of inflammatory mediators in systemic circulation.

Gut microbiome manipulation, for example through the use of probiotic and prebiotic supplements, has shown some promise in the treatment of IBS. However, the research in this area is still in its infancy, and it remains unclear what type of intervention that is the preferred choice in cases of IBS.

Several studies have investigated how the use of probiotic supplements containing Bifidobacteria and Lactobacilli affect the clinical outcome of patients with IBS. However, to date, no studies have assessed whether fermented vegetables, a "natural" source of probiotic bacteria such as Lactobacillus plantarum, are useful in the treatment of IBS.

ELIGIBILITY:
Inclusion Criteria:

Rome III criteria (Criteria fulfilled for the last 6 months with symptom onset at least 3 months prior to diagnosis):

Recurrent abdominal pain or discomfort at least 3 days/month in the last 3 months associated with two or more of the following:

1. Improvement with defecation
2. Onset associated with a change in frequency of stool
3. Onset associated with a change in form (appearance) of stool

Exclusion Criteria:

* Psychiatric disorder
* Metabolic disease
* Chronic infection
* Organic gastrointestinal disorder
* Pregnancy
* Breastfeeding

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-09; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
IBS Symptom Severity Scale (IBS-SSS). | Change from day 0 to day 42

SECONDARY OUTCOMES:
Body weight | Change from day 0 to day 42
Fecal microbiome diversity | Change from day 0 to day 42
  16S rRNA gene sequences (prokaryotes)
The Quality of Life Scale (QOLS) | Change from day 0 to day 42

CONTACTS AND LOCATIONS:
Locations (1):
- Volvat Medisinske Senter, Majorstuen, Oslo, Norway